CLINICAL TRIAL: NCT03092102
Title: A Phase I, Double-blind, Placebo-controlled, Single and Multiple Oral Dose, Safety, Tolerability and Pharmacokinetic Study of HEC585 in Healthy Male and Female Subjects
Brief Title: The Safety, Tolerability and Pharmacokinetic Study of HEC585 in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCD-DHEC585-16-001
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- A single dose HEC585（A1） (Experimental): Drug: HEC585 Capsule
  Drug: HEC585-matching placebo Capsule
  Interventions: Drug: HEC585
- A single dose HEC585（A2） (Experimental): Drug: HEC585 Capsule
  Drug: HEC585-matching placebo Capsule
  Interventions: Drug: HEC585
- A single dose HEC585/FE（A3） (Experimental): Drug: HEC585 Capsule
  Drug: HEC585-matching placebo Capsule
  Treatment Period 1：No food prior to dosing；Treatment Period 2：High-fat meal prior to dosing
  Interventions: Drug: HEC585
- A single dose HEC585（A4） (Experimental): Drug: HEC585 Capsule
  Drug: HEC585-matching placebo Capsule
  Interventions: Drug: HEC585
- A single dose HEC585（A5） (Experimental): Drug: HEC585 Capsule
  Drug: HEC585-matching placebo Capsule
  Interventions: Drug: HEC585
- A single dose HEC585（A6） (Experimental): Drug: HEC585 Capsule
  Drug: HEC585-matching placebo Capsule
  Interventions: Drug: HEC585
- A single dose HEC585（A7） (Experimental): Drug: HEC585 Capsule
  Drug: HEC585-matching placebo Capsule
  Interventions: Drug: HEC585
- A single dose HEC585（A8） (Experimental): Drug: HEC585 Capsule
  Drug: HEC585-matching placebo Capsule
  Interventions: Drug: HEC585
- Multiple doses HEC585（B1） (Experimental): Drug: HEC585 Capsule
  Drug: HEC585-matching placebo Capsule
  Interventions: Drug: HEC585
- Multiple doses HEC585（B2） (Experimental): Drug: HEC585 Capsule
  Drug: HEC585-matching placebo Capsule
  Interventions: Drug: HEC585
- Multiple doses HEC585（B3） (Experimental): Drug: HEC585 Capsule
  Drug: HEC585-matching placebo Capsule
  Interventions: Drug: HEC585
- Multiple doses HEC585（B4） (Experimental): Drug: HEC585 Capsule
  Drug: HEC585-matching placebo Capsule
  Interventions: Drug: HEC585
- Multiple doses HEC585（B5） (Experimental): Drug: HEC585 Capsule
  Drug: HEC585-matching placebo Capsule
  Interventions: Drug: HEC585
- Multiple doses HEC585（B6） (Experimental): Drug: HEC585 Capsule
  Drug: HEC585-matching placebo Capsule
  Interventions: Drug: HEC585

INTERVENTIONS:
Drug: HEC585 — HEC585, a pyrimidone compound, is structurally related to pirfenidone, a pyridine compound.

SUMMARY:
The Safety, Tolerability and Pharmacokinetic Study of idiopathic pulmonary fibrosis treatment drug HEC585 in Healthy Male and Female Subjects

DETAILED DESCRIPTION:
This will be a double-blind, placebo-controlled, single, and multiple oral dose study conducted in 2 parts.

Part A will comprise a single-dose, sequential-group study incorporating a food effect evaluation. Up to 48 subjects will be studied in up to 6 groups (Groups A1 to A6), with each group consisting of 8 subjects. Each subject will participate in 1 treatment period only and reside at the clinical research unit (CRU) from Day -1 (the day before dosing) to Day 7 (144 hours postdose), except for Group A3, which will participate in a second treatment period for a food effect evaluation. Each subject in Group A3 will participate in 2 treatment periods separated by a minimum of 7 days. Dosing of subjects in the fed state in Group A3 can commence after review of the safety data from Group A4.

Part B will comprise a multiple-dose, sequential-group study. Up to 36 subjects will be studied in up to 3 groups (Groups B1 to B3), with each group consisting of 12 subjects. Part B of the study may start after completion of Group A5, at a dose equal or less than given in Groups A1 to A3.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, of any race, between 18 and 60 years of age, inclusive, at Screening.
2. Body mass index between 18.0 and 32.0 kg/m2, inclusive, at Screening.
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, Gilbert's syndrome] is not acceptable) at Screening and/or Check-in as assessed by the Investigator (or designee).
4. Females will be nonpregnant and nonlactating. Females of childbearing potential and male subjects will agree to use contraception.
5. Able to comprehend and willing to sign an informed consent form (ICF) and to abide by the study restrictions.

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
3. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).
4. History of alcoholism or drug/chemical abuse within 2 years prior to Check-in.
5. Alcohol consumption of > 21 units per week for males and > 14 units for females. One unit of alcohol equals 12 oz (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL wine), or a positive alcohol breath test at Check-in.
6. Positive urine drugs of abuse screen including cotinine at Screening or Check-in.
7. Positive hepatitis B surface antigen, hepatitis C virus antibody and/or positive human immunodeficiency virus (HIV) test (Appendix 3).
8. Absolute lymphocyte count below the lower limit of normal which can be confirmed by repeat.
9. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days or 5 half-lives (if known), whichever is longer, prior to Check-in.
10. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's Wort, within 30 days prior to Check-in, unless deemed acceptable by the Investigator (or designee). Strong CYP3A inhibitors and inducers should be avoided.
11. Use or intend to use any prescription medications/products, within 14 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
12. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within 7 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
13. Use of tobacco- or nicotine-containing products within 3 months prior to Check-in.
14. Consumption of foods and beverages containing poppy seeds, grapefruit, or Seville oranges within 7 days prior to Check-in, consumption of caffeine-containing foods and beverages within 72 hours prior to Check-in, or consumption of alcohol within 48 hours prior to Check-in.
15. Receipt of blood products within 2 months prior to Check-in.
16. Donation of blood from 56 days prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.
17. Poor peripheral venous access.
18. Have previously completed or withdrawn from this study, and have previously received the investigational product.
19. Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Cmax | Predose, and 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144,and 216 h
  Geometric Mean of Maximum Observed Plasma Concentration of HEC585
(AUC0-∞） | Predose, and 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120,144,and 216 h
  area under the plasma concentration-time curve (AUC) from time zero to infinity
tmax | Predose, and 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144,and 216 h
  time of the maximum observed plasma concentration
Vz/F | Predose, and 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120,144,and 216 h
  apparent volume of distribution
t½ | Predose, and 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144,and 216 h
  apparent terminal elimination half-life
CL/F | Predose, and 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144,and 216 h
  apparent oral clearance

SECONDARY OUTCOMES:
Adverse event | From baseline to 7 days
  To assess the safety and tolerability of 7 days therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit, Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No